CLINICAL TRIAL: NCT02304848
Title: Effects of Deep Brain Stimulation (DBS) Frequency on Neural Synchrony
Acronym: DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, Dr, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60130
Record Dates: First submitted 2014-08-06; First posted 2014-12-02 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; DBS; Deep Brain Stimulation; Subthalamic Nucleus
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

ARMS (1):
- DBS (Deep Brain Stimulation) (Experimental): DBS ( Deep Brain Stimulation) ( both high and low frequency deep brain stimulation will be applied to the subthalamic nucleus)
  Interventions: Other: DBS (Deep Brain Stimulation)

INTERVENTIONS:
Other: DBS (Deep Brain Stimulation) — Applying low frequency and high frequency deep brain stimulation to subthalamic nucleus.

SUMMARY:
The purpose of this study is to evaluate the effects of low frequency deep brain stimulation on subthalamic nucleus neural synchrony. Low frequency stimulation does not improve the cardinal motor signs of Parkinson's disease, and may be beneficial only for gait and speech. This study will provide insight into what the effects of low frequency stimulation are on neural synchrony.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic Parkinson's disease, with bilateral symptoms at Hoehn and Yahr Stage greater than or equal to II.
* Documented improvement in motor signs on versus off dopaminergic medication, with a change in the Unified Parkinson's Disease Rating Scale motor (UPDRS III) score of >= 30% off to on medication.
* The presence of complications of medication such as wearing off signs, fluctuating responses and/or dyskinesias, and/or medication refractory tremor, and/or impairment in the quality of life on or off medication due to these factors.
* Subjects should be on stable doses of medications, which should remain unchanged until the DBS system is activated. After the DBS system is optimized (during which time the overall medication dose may be reduced to avoid discomfort and complications such as dyskinesias) the medication dose should remain unchanged, if possible, for the duration of the study.
* Treatment with carbidopa/levodopa, and with a dopamine agonist at the maximal tolerated doses as determined by a movement disorders neurologist.
* Age > 18

Exclusion Criteria:

* Subjects with significant cognitive impairment and/or dementia as determined by a standardized neuropsychological battery.
* Subjects with clinically active depression, defined according to the Diagnostic and Statistical manual of Mental Disorders, Fourth Edition (DSM-IV) criteria and as scored on a validated depression assessment scale.
* Subjects with very advanced Parkinson's disease, Hoehn and Yahr stage 5 on medication (non-ambulatory).
* Age > 80.
* Subjects with an implanted electronic device such as a neurostimulator, cardiac pacemaker/defibrillator or medication pump.
* Subjects, who are pregnant, are capable of becoming pregnant, or who are breast feeding.
* Patients with cortical atrophy out of proportion to age or focal brain lesions that could indicate a non-idiopathic movement disorder as determined by MRI
* Subjects having a major comorbidity increasing the risk of surgery (prior stroke, severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin).
* Subjects having any prior intracranial surgery.
* Subjects with a history of seizures.
* Subjects, who are immunocompromised.
* Subjects with an active infection.
* Subjects, who require diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS) to treat a chronic condition.
* Subjects, who have an inability to comply with study follow-up visits.
* Subjects, who are unable to understand or sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-10; Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Low frequency stimulation versus no stimulation | 3 years
  The changes in neuronal oscillations, measured in power (dB/Hz) and frequency (Hz), that are significantly different between periods of low frequency stimulation and periods of no stimulation - during rest - in people with Parkinson's disease off medications.

SECONDARY OUTCOMES:
Low frequency stimulation versus high frequency stimulation | 3 years
  To determine if the effects of low frequency stimulation are due to using a lower total power delivered than normal therapeutic high frequency stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MD, MSE, FAAN, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Derived] O'Day J, Syrkin-Nikolau J, Anidi C, Kidzinski L, Delp S, Bronte-Stewart H. The turning and barrier course reveals gait parameters for detecting freezing of gait and measuring the efficacy of deep brain stimulation. PLoS One. 2020 Apr 29;15(4):e0231984. doi: 10.1371/journal.pone.0231984. eCollection 2020. PMID 32348346